CLINICAL TRIAL: NCT02703688
Title: Environmental Influences on Early Childhood Obesity: The Healthy Homes Study
Brief Title: Environmental Influences on Early Childhood Obesity
Acronym: HHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-1975; K23DK087826 (NIH)
Record Dates: First submitted 2016-02-22; First posted 2016-03-09 (Estimated); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Homes (Experimental): Behavioral Intervention
  Interventions: Behavioral: Healthy Homes
- Usual Care (Active Comparator): Counseling session delivered by pediatrician
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Healthy Homes — The Healthy Homes Behavioral Intervention (HHBI) will be delivered during 8 sessions over 10 weeks using home visitations. The first 6 sessions occur weekly and provide education about healthy dietary intake including caloric recommendations for preschool aged children, healthy sleep goals, active play and screen time limits, and family routines and organization. Each session will include a parent-child interaction component to teach child behavior management skills related to intervention goals. Two final sessions occur every other week to provide problem solving and planning for maintenance of treatment effects.
  Arms: Healthy Homes
Other: Usual Care — A pediatrician with experience delivering weight management treatment to children will deliver a single session, 1-hour treatment to families. Content to be delivered during the session will include lifestyle recommendations currently recommended by the AAP.
  Arms: Usual Care

SUMMARY:
Few treatments have been developed for young children with obesity from diverse backgrounds. The present study will develop and test an intervention designed to improve preschool obesity in Latino children. The intervention will focus on improving eating, activity, and sleep behaviors and the home environment for improved weight status.

DETAILED DESCRIPTION:
Children from low income families of minority status are at greater risk for development of obesity. There are no known existing treatments for pediatric obesity that focus on improving parental behaviors and the home food and activity environment. The objective of this study will be to address this limitation by developing and testing a novel treatment for low-income minority families. The objective will be attained by testing the following hypothesis: A parent-focused, home-based treatment aimed at improving parental feeding behaviors, child exposure to fruits and vegetables, and the home food and activity environment will result in significantly greater decrease in percent overweight / obesity compared to recommended practice. The hypothesis will be tested by using the approach of a pilot randomized control trial (RCT). The rationale for this aim is that success of the planned research will derive a treatment package that will provide the basis for the RCT. The planned research is expected to show the level of impact of changing parental feeding behaviors and the home environment on childhood overweight / obesity.

ELIGIBILITY:
Inclusion Criteria:

1. mothers will identify themselves as being Latino
2. obese preschool children will be required to have a BMI percentile at or above the 95th percentile, based on sex specific, BMI-for-age population referenced growth charts
3. participating children will be required to have at least one primary caregiver who is English-speaking as their primary language and live within 50 miles of the UCD for the initial treatment development phase (n=3) and at least one family who is Spanish speaking (n=1). However, all families participating in the randomized portion can also be exclusively Spanish speaking.

Exclusion Criteria:

1. Children with medical conditions known to promote obesity will be excluded along with individuals involved with a weight-control program or those taking appetite-affecting medications
2. Children who are greater than 100% overweight
3. Children will be excluded who have a reported disability, illness, or disorder that would significantly affect diet or activity behaviors
4. children identified by parents with significant food allergies
5. involvement with Stage II, structured weight management for obesity.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 129 (Actual)
Dates: Start 2011-09-15 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2014-03-31 (Actual)

PRIMARY OUTCOMES:
Change in BMI | Baseline, 2.5 months, 12 months
  BMI and % over the 95th percentile will be determined using scales

SECONDARY OUTCOMES:
Change in Caregiver's Feeding Styles Questionnaire | Baseline, 2.5 months, 12 months
  Change in type of parental feeding style over time
Change in Child caloric intake | Baseline, 2.5 months, 12 months
  24 hour dietary recall will identify average daily caloric intake
Change in Sleep duration | Baseline, 2.5 months, 12 months
  Accelerometer will be used to determine objective estimates of sleep duration
Change in Home sleep environment | Baseline, 2.5 months, 12 months
  change in sleeping environment characteristics that promote healthy sleep
Change in Home food environment | Baseline, 2.5 months, 12 months
  change in home food environment characteristics that promote healthy food intake.

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Boles, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided